CLINICAL TRIAL: NCT05439538
Title: Serum Neutrophil Gelatinase-associated Lipocalin (NGAL) as a Predictor of Renal Injury in Patients With Multiple Myeloma
Brief Title: Serum NGAL IN Patients With Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ehab A. Abdelmenam, Principal Investigator, Assiut University
Other Study IDs: NGAL IN MM
Record Dates: First submitted 2022-06-23; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma(MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SERUM NGAL — Study the sensitivity and the specificity of serum NGAL to detect AKI in myeloma

SUMMARY:
The aim of this study was to evaluate SERUM neutrophil gelatinase-associated lipocalin, emerging indicator of tubular damage and examine their relationship with established measures of renal function (serum creatinine, and estimated glomerular filtration rate, eGFR) among MM patients with and without renal impairment (RI), and at various stages of MM progression.

DETAILED DESCRIPTION:
Multiple myeloma (MM), Being one of the most common hematologic malignancies, particularly in the elderly patient, MM represents a devastating disease that occurs due to uncontrolled proliferation of a plasma cell in bone marrow , MM Presents itself with characteristic features of organ involvement: bone lesions, anemia, renal insufficiency, infections, hypercalcemia and specific malignancy biomarkers (plasma cell clonality ≥60%, involved to uninvolved serum free light chains (FLCs) ≥100 and >1 focal lesion on magnetic resonance imaging) . Additionally , Evidence of clonal plasma cell percentage of ≥10% in bone marrow or biopsy-proven plasmacytoma is necessary to define a case of MM .

MM is the second most commonly diagnosed hematological neoplasm, with an incidence rate of 5.3 per 100 000 individuals ,its incidence in Egypt 1.5 per 100 000 individuals Early mortality may not only be associated with disease progression, but also with concomitant organ involvement (i.e., renal failure) and therapy side-effects (i.e., infections) .

Production of monoclonal paraproteins, immunoglobulins (MIg) or free light chains (FLCs), is a characteristic feature of myeloma that is tied to its clinical manifestations,Although non-functional, paraproteins may be produced in excess, which alongside their physicochemical properties may precipitate the formation of lesions in vasculature and variably affect organ function. Owing to the differences between individual clones and associated MIg, kidney pathology is highly heterogeneous, with renal tubular injury associated with light chain cast nephropathy as the dominant presentation .

Renal impairment (RI) is one of the most common complications of symptomatic MM(close to one fourth of patients at the time of diagnosis). RI, defined as a serum creatinine (sCr) level > 2 mg/dL, is one of the diagnostic criteria of symptomatic MM, and it constitutes 1 of the 4 "CRAB" features (calcium level elevation, renal impairment, anemia, and bone lesions) that indicate myeloma-related organ dysfunction .. RI can carry a poor prognosis, particularly if renal function does not recover , Irreversible renal failure is less frequent, but may be present in up to 8% of patients .

The use of novel antimyeloma agents such as proteasome inhibitors (PIs) and immunomodulatory drugs (IMiDs) as well as the improvement in supportive care has resulted in a substantial increase in patient survival. However, RI reversibility is still closely associated with MM prognosis. The persistence of severe RI is associated with significant morbidity and mortality, and remains one of the factors associated with early death, Effective anti-MM therapy and supportive care can restore renal function in several patients, Therefore, earlier recognition of disease, including its end-organ manifestations, is necessary for timely initiation and optimization of therapy but we lack biomarkers that could predict renal outcomes . Renal insufficiency is considered reversible in about 50% of cases in some reports .

Around 10% of them require haemodialysis, with a negative impact on prognosis. In addition, half of MM patients will present with at least one episode of acute kidney injury during the course of their disease. Acute kidney injury mostly reflects high tumour burden disease .

The standard assessment of renal function in patients with MM includes the measurement of sCr concentration, creatinine clearance (CrCl), blood urea nitrogen, and Estimated Glomerular Filtration Rate (eGFR), as calculated using the EPI equation. However, sCr is primarily a marker of glomerular filtration and reliant on a number of non-renal factors(comorbidity, muscle mass, medication, age), if GFR is not significantly reduced, sCr is an insensitive and late marker in the diagnosis of renal tubular injury. Novel biomarkers that will aid in predicting renal injury and chronic kidney disease development are of high interest and very early and sensitive markers .

AKI classified according to the Acute Kidney Injury Network (AKIN) classification into three stages: stage 1 Increase in serum creatinine of ≥0.3 mg/dL, stage 2 Increase in serum creatinine to 200 to 300% baseline ,stage 3 Increase in serum creatinine to >300% baseline .

One of the most promising and earliest biomarkers of kidney injury is neutrophil gelatinase-associated lipocalin (NGAL) (lipocalin 2 [LCN2]). NGAL is a lipocalin iron-carrying protein of 25 KDa expressed at low levels in several human tissues, including the kidney(16). NGAL is one of the earliest and most robust markers of acute kidney injury), reflects renal function more accurately than creatinine and correlates with both tumor burden and renal function in MM, The advantage of NGAL over conventional biomarkers of RI such as sCr and serum urea nitrogen is that the levels often increase long before any changes in sCr or urea nitrogen or urine output occur. Therefore, NGAL may also be an early, sensitive marker of RI in patients with MM .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) with SMM or overt multiple myeloma (MM will be confirmed based on the WHO diagnostic criteria; the presence of at least 10% plasma cells in bone marrow biopsies, presence of momoclonal protein in serum and /or urine and one of the following disorders (CRAB): hypercalcemia, renal failure, anemia, or lytic bone lesions).

Exclusion Criteria:

* ( other causes affect NAGAL level )

  1. Patients with other plasma cell disorders (eg. Waldenstrom macroglobulinuria, MGUS, amyloidosis )
  2. Recent active infection;
  3. History of hepatitis B, C, or HIV
  4. Neoplasms other than myeloma

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — adult MM patients more than 18 years
Study Population: Patients will be recruited during admission and visits to Clinical Hematology Unit and outpatients clinic, Assiut university hospital, from October 2022 to October 2023.
  Sample size is 60 patients diagnosed MM with or without renal impairment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
serum Neutrophil Gelatinase-associated Lipocalin in patients with multiple myeloma | baseline to 3 months
  Role of serum Neutrophil Gelatinase-associated Lipocalin in early detection of renal impairment in patients with multiple myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Essam Abdel Monem El-beih,, professor, Study Director — Assiut Univ

REFERENCES:
- [Background] Turesson I, Bjorkholm M, Blimark CH, Kristinsson S, Velez R, Landgren O. Rapidly changing myeloma epidemiology in the general population: Increased incidence, older patients, and longer survival. Eur J Haematol. 2018 Apr 20:10.1111/ejh.13083. doi: 10.1111/ejh.13083. Online ahead of print. PMID 29676004
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Ludwig H, Novis Durie S, Meckl A, Hinke A, Durie B. Multiple Myeloma Incidence and Mortality Around the Globe; Interrelations Between Health Access and Quality, Economic Resources, and Patient Empowerment. Oncologist. 2020 Sep;25(9):e1406-e1413. doi: 10.1634/theoncologist.2020-0141. Epub 2020 May 7. PMID 32335971
- [Background] Mohty M, Cavo M, Fink L, Gonzalez-McQuire S, Leleu H, Mateos MV, Raab MS, Schoen P, Yong K. Understanding mortality in multiple myeloma: Findings of a European retrospective chart review. Eur J Haematol. 2019 Aug;103(2):107-115. doi: 10.1111/ejh.13264. Epub 2019 Jun 18. PMID 31112311
- [Background] Rafae A, Malik MN, Abu Zar M, Durer S, Durer C. An Overview of Light Chain Multiple Myeloma: Clinical Characteristics and Rarities, Management Strategies, and Disease Monitoring. Cureus. 2018 Aug 15;10(8):e3148. doi: 10.7759/cureus.3148. PMID 30345204
- [Background] Gonsalves WI, Milani P, Derudas D, Buadi FK. The next generation of novel therapies for the management of relapsed multiple myeloma. Future Oncol. 2017 Jan;13(1):63-75. doi: 10.2217/fon-2016-0200. Epub 2016 Aug 11. PMID 27513456
- [Background] Evison F, Sangha J, Yadav P, Aung YS, Sharif A, Pinney JA, Drayson MT, Cook M, Cockwell P. A population-based study of the impact of dialysis on mortality in multiple myeloma. Br J Haematol. 2018 Feb;180(4):588-591. doi: 10.1111/bjh.14394. Epub 2016 Oct 21. No abstract available. PMID 27766629
- [Background] Clerico A, Galli C, Fortunato A, Ronco C. Neutrophil gelatinase-associated lipocalin (NGAL) as biomarker of acute kidney injury: a review of the laboratory characteristics and clinical evidences. Clin Chem Lab Med. 2012 Feb 15;50(9):1505-17. doi: 10.1515/cclm-2011-0814. PMID 22962216